CLINICAL TRIAL: NCT05063292
Title: Effect of Prewarming On Skin Temperature Changes After Spinal Anesthesia in Transurethral Resection of The Bladder
Brief Title: Effect of Prewarming On Skin Temperature Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, NEGIN NAYEBI, MD, Anesthesiology Resident, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NeginIzmirBozyaka
Record Dates: First submitted 2021-08-31; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Spinal Anesthesia; Hypothermia Following Anesthesia; Prewarming; Core Temperature; Urological Cancer
Keywords: hypothermia; peripheral temperature; spinal anesthesia; forced-air warming
MeSH Terms: conditions — Urologic Neoplasms; Hypothermia

STUDY DESIGN:
Intervention Model Description: The study covers 2 groups. Group I will be covered with warmed double layered cotton cloth. Group II will be covered with air forced blanket.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients covered with a 41 centigrade degrees double layered cotton cloth
- Prewarmed group (Experimental): Patients receive active prewarming with an air forced blanket ( full body blanket) 30 minutes prior to the operation
  Interventions: Procedure: Patients in Group II will receive active prewarming with an air forced blanket (full body blanket) 30 minutes prior to the operation

INTERVENTIONS:
Procedure: Patients in Group II will receive active prewarming with an air forced blanket (full body blanket) 30 minutes prior to the operation — Core temperature and 4-points skin temperatures measurements will be recorded all over the operation. Patients will be delivered 2 Litre/minute oxygen with a nasal cannula.Iv hydration will be continued by room temperatured balanced electrolyte solution with an infusion rate of 2mL/kg/hr. Spinal anesthesia will be applied at the level of L3-L4 by a 25 Gauge Quincke needle with a dose of 12.5-15 mg hyperbaric bupivacaine in the sitting position.
  Arms: Prewarmed group

SUMMARY:
In this randomized prospective single-blind study,American Society of Anesthesiologists physical status classification system ( ASA )I-II-III patients aged 50-80 years undergoing transurethral bladder resection will be randomly divided into two groups. First group will be covered with 41 centigrade degrees double layered cotton cloth. Second group will receive active prewarming. Core temperature of all patients will be monitorized via tympanic membrane. Skin temperature will be monitorized from 4 different body areas. Spinal anesthesia will be applied at the level of L3-L4 by a 25 Gauge quincke needle with a dose of 12.5-15 mg hyperbaric bupivacaine. Pinprick test will be used for sensorial block assessment. T10 sensorial block will be our goal. Hemodynamic parameters will be recorded. Skin temperature will be monitorized before and after spinal anesthesia and changes will be recorded. Operation time, amount and temperature of irrigation fluids, transfusion requirement, discharge time from postoperative care unit will also be recorded. Shivering score and thermal comfort scale will be used. The two groups will be compared for the temperature changes.

DETAILED DESCRIPTION:
In this prospective single-blind study, patients will be divided into 2 groups with computer-based randomization technique. All patients will have a fasting time of 2 hours for clear fluid and 6 hours for solid food. Patients will be taken to the premedication room before the operation. Written and verbal approval will be taken from all patients. Tympanic membrane will be used for core temperature measurement by Citizen ear thermometer,every 15 minutes.Adult skin temperature probe will be used for continuous peripheral temperature measurement from four different body areas (T1:Cervical7 (C7) dermatome, T2:C6 dermatome T3:Lumbar 5( L5 )dermatome, T4: L4 dermatome). The two groups will have an infusion of balanced electrolyte solution with a rate of 8 Mililitre/Kilogram/ hour(mL/kg/hour). Patients in Group I will be covered with a 41 centigrade degrees double layered cotton clothes. Patients in Group II will receive active prewarming with a forced-air warming blanket (WarmCare full body blanket) 30 minutes prior to the operation. 0.1 mg/kg intravenous (iv) midazolam hydrochloride will be administered for premedication. Patients will be transferred to operating room, covered with warmed double layered cotton clothes. Standard monitoring (pulse oximetry, noninvasive blood pressure, electrocardiography) will be applied to the patients. Core temperature and 4-points skin temperature measurements will be recorded. Patients will be delivered 2 Liter/minute oxygen with a nasal cannula. Iv hydration will be continued by room temperature balanced electrolyte solution with an infusion rate of 2mililiter/kilogram/hour. Spinal anesthesia will be applied at the level of L3-L4 by a 25 Gauge Quincke needle with a dose of 12.5-15 mg hyperbaric bupivacaine in the sitting position. Then patients will be taken supine position. Hemodynamic measurements will be continued. Core temperature measurements will be done every 15 minutes. Peripheral skin temperature measurements will be continuous. 1st, 2nd ,3rd,4th ,5th ,6th, 7th, 8th, 9th and 10th minutes and every 5 minutes measurements will be recorded during the operation. Pinprick test will be used for sensorial block assessment. T10 sensorial block will be our goal. The time for adequate sensorial block (T10) will be recorded. The patients will be repositioned (lithotomy) before the beginning of surgery. 5 mg iv ephedrine and 0.5 mg iv atropine will be administered when the blood pressure will be %80 of the baseline pressure and heart rate. Operating time, amount and temperature of irrigation fluids, transfusion requirement will be recorded. All patients will be transferred to post anesthesia care unit (PACU). Core temperature measurements will be continued every 15 minutes at PACU. Shivering scale and thermal comfort scale will be used during and after the operation. 25 mg iv meperidine will be administered when the patient's shivering score will be more than 3. Length of PACU stay will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III
* 50-80 years old
* Patients scheduled for transurethral baldder resection

Exclusion Criteria:

* Female gender
* Uncoordinated patients
* Have coagulopathy,
* Known allergies to drugs to be used,
* Patients diagnosed with severe hypovolemia
* Skin infection at the injection site.
* Body mass index greater than 35m2/kg
* patients with severe endocrinological disease
* Patients with cardiovascular diseases
* patients with severe aortic stenosis or severe mitral stenosis
* patients with increased intracranial pressure

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients scheduled for transurethral bladder resection
Enrollment: 60 (Estimated)
Dates: Start 2021-10-05 (Estimated); Primary Completion 2021-11-10 (Estimated); Study Completion 2021-11-18 (Estimated)

PRIMARY OUTCOMES:
peripheral skin temperature at ( F0) | just after spinal anesthesia done
  F0 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature at( S0) | just after spinal anesthesia done
  S0 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature( T0) | just after spinal anesthesia done
  T0 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( M0) | just after spinal anesthesia done
  M0 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( F1) | 60 seconds after spinal anesthesia done
  F1will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F2) | 120 seconds after spinal anesthesia done
  F2 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F3) | 180 seconds after spinal anesthesia done
  F3 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F4) | 4 minute after spinal anesthesia done
  F4 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F5) | 5 minute after spinal anesthesia done
  F5 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F6) | 6 minute after spinal anesthesia done
  F6 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F7) | 7 minute after spinal anesthesia done
  F7 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F8) | 8 minute after spinal anesthesia done
  F8 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F9) | 9 minute after spinal anesthesia done
  F9 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F10) | 10 minute after spinal anesthesia done
  F10 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F15) | 15 minute after spinal anesthesia done
  F15 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F20) | 20 minute after spinal anesthesia done
  F20 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F25) | 25 minute after spinal anesthesia done
  F25 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F30) | 30 minute after spinal anesthesia done
  F30 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F35) | 35 minute after spinal anesthesia done
  F35 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F40) | 40 minute after spinal anesthesia done
  F40 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F45) | 45 minute after spinal anesthesia done
  F45 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F50) | 50 minute after spinal anesthesia done
  F50 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F55) | 55 minute after spinal anesthesia done
  F55 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature( F60) | 60 minute after spinal anesthesia done
  F60 will be defined as temperature which measured at C7 dermatome from palmar side of the 3rd finger with adult skin probe
peripheral skin temperature at( S1) | 60 seconds after spinal anesthesia done
  S1 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S2) | 120 seconds after spinal anesthesia done
  S2 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S3) | 180 seconds after spinal anesthesia done
  S3 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S4) | 4 minute after spinal anesthesia done
  S4 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S5) | 5 minute after spinal anesthesia done
  S5 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S6) | 6 minute after spinal anesthesia done
  S6 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S7) | 7 minute after spinal anesthesia done
  S7 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S8) | 8 minute after spinal anesthesia done
  S8 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S9) | 9 minute after spinal anesthesia done
  S9 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S10) | 10 minute after spinal anesthesia done
  S10 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S15) | 15 minute after spinal anesthesia done
  S15 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S20) | 20 minute after spinal anesthesia done
  S20 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S25) | 25 minute after spinal anesthesia done
  S25 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S30) | 30 minute after spinal anesthesia done
  S30 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S35) | 35 minute after spinal anesthesia done
  S35 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S40) | 40 minute after spinal anesthesia done
  S40 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S45) | 45 minute after spinal anesthesia done
  S45 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S50) | 50 minute after spinal anesthesia done
  S50 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S55) | 55 minute after spinal anesthesia done
  S55 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature at( S60) | 60 minute after spinal anesthesia done
  S60 will be defined as temperature which measured at C6 dermatome from ventral side of styloid process with adult skin probe
peripheral skin temperature( T1) | 60 seconds after spinal anesthesia done
  T1 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T2) | 120 seconds after spinal anesthesia done
  T2 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T3) | 180 seconds after spinal anesthesia done
  T3 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T4) | 4 minute after spinal anesthesia done
  T4 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T5) | 5 minute after spinal anesthesia done
  T5 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T6) | 6 minute after spinal anesthesia done
  T6 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T7) | 7 minute after spinal anesthesia done
  T7 will be defined as temperature which measured at L5 deramatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T8) | 8 minute after spinal anesthesia done
  T8 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T9) | 9 minute after spinal anesthesia done
  T9 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T10) | 10 minute after spinal anesthesia done
  T10 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T15) | 15 minute after spinal anesthesia done
  T15 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T20) | 20 minute after spinal anesthesia done
  T20 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T25) | 25 minute after spinal anesthesia done
  T25 will be defined as temperature which measured L5 dermatome at plantar side of 1st toe with adult skin probe
peripheral skin temperature( T30) | 30 minute after spinal anesthesia done
  T30 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T35) | 35 minute after spinal anesthesia done
  T35 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T40) | 40 minute after spinal anesthesia done
  T40 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T45) | 45 minute after spinal anesthesia done
  T45will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T50) | 50 minute after spinal anesthesia done
  T50 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T55) | 55 minute after spinal anesthesia done
  T55 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( T60) | 60 minute after spinal anesthesia done
  T60 will be defined as temperature which measured at L5 dermatome plantar side of 1st toe with adult skin probe
peripheral skin temperature( M1) | 60 seconds after spinal anesthesia done
  M1 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M2) | 120 seconds after spinal anesthesia done
  M2 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M3) | 180 seconds after spinal anesthesia done
  M3 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M4) | 4 minute after spinal anesthesia done
  M4 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M5) | 5 minute after spinal anesthesia done
  M5 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M6) | 6 minute after spinal anesthesia done
  M6 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M7) | 7 minute after spinal anesthesia done
  M7 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M8) | 8 minute after spinal anesthesia done
  M8 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M9) | 9 minute after spinal anesthesia done
  M9 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M10) | 10 minute after spinal anesthesia done
  M10 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M15) | 15 minute after spinal anesthesia done
  M15 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M20) | 20 minute after spinal anesthesia done
  M20 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M25) | 25 minute after spinal anesthesia done
  M25 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M30) | 30 minute after spinal anesthesia done
  M30 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M35) | 35 minute after spinal anesthesia done
  M35 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M40) | 40 minute after spinal anesthesia done
  M40 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M45) | 45 minute after spinal anesthesia done
  M45 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M50) | 50 minute after spinal anesthesia done
  M50 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M55) | 55 minute after spinal anesthesia done
  M55 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe
peripheral skin temperature( M60) | 60 minute after spinal anesthesia done
  M60 will be defined as temperature which measured at L4 dermatome above the medial malleolus with adult skin probe

SECONDARY OUTCOMES:
core tympanic membrane temperature (C0) | just before spinal anesthesia done
  centigrade degree , Timpanic membrane will be used for core temperature measurement by Citizen ear thermometer, CTD504,
core tympanic membrane temperature(C1) | 15 minute after spinal anesthesia done
  centigrade degree , Tympanic membrane will be used for core temperature measurement by Citizen ear thermometer, CTD504,
core tympanic membrane temperature(C2) | 30 minute after spinal anesthesia done
  centigrade degree , Tympanic membrane will be used for core temperature measurement by Citizen ear thermometer, CTD504,
core tympanic membrane temperature(C3) | 45 minute after spinal anesthesia done
  centigrade degree , Tympanic membrane will be used for core temperature measurement by Citizen ear thermometer, CTD504,
core tympanic membrane temperature(C4) | 60 minute after spinal anesthesia done
  centigrade degree , Tympanic membrane will be used for core temperature measurement by Citizen ear thermometer, CTD504,
thermal comfort scale | Immediately after the surgery
  thermal comfort will be rated on a 100mm visual analog scale (VAS),with zero indicating intense cold and 100mm representing intense heat
shivering score(h0) | just before spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body
shivering score(h1) | 15 minute after spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body
shivering score(h2) | 30 minute after spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body
shivering score(h3) | 45 minute after spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body
shivering score(h4) | 60 minute after spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body
shivering score(h5) | 75 minute after spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body
shivering score(h6) | 90 minute after spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body
shivering score(h7) | 105 minute after spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body
shivering score(h8) | 120 minute after spinal anesthesia done
  0: no shivering 1:piloerection or peripheral vasoconstriction but no visible shivering 2: muscular activity in only one muscle group 3:muscular activity in more then one muscle group but not generalized shivering 4:shivering involving the whole body

CONTACTS AND LOCATIONS:
Overall Officials: Halide Hande Şahinkaya, Specialist, Study Chair — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Bozyaka Training and Research Hospital, Izmir, Karabağlar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hermanns H, Werdehausen R, Hollmann MW, Stevens MF. Assessment of skin temperature during regional anaesthesia-What the anaesthesiologist should know. Acta Anaesthesiol Scand. 2018 Oct;62(9):1280-1289. doi: 10.1111/aas.13176. Epub 2018 Jun 25. PMID 29938773
- [Background] Jun JH, Chung MH, Kim EM, Jun IJ, Kim JH, Hyeon JS, Lee MH, Lee HS, Choi EM. Effect of pre-warming on perioperative hypothermia during holmium laser enucleation of the prostate under spinal anesthesia: a prospective randomized controlled trial. BMC Anesthesiol. 2018 Dec 22;18(1):201. doi: 10.1186/s12871-018-0668-4. PMID 30579334
- [Background] Fradkin AJ, Zazryn TR, Smoliga JM. Effects of warming-up on physical performance: a systematic review with meta-analysis. J Strength Cond Res. 2010 Jan;24(1):140-8. doi: 10.1519/JSC.0b013e3181c643a0. PMID 19996770
- [Background] Frank SM, El-Rahmany HK, Tran KM, Vu B, Raja SN. Comparison of lower extremity cutaneous temperature changes in patients receiving lumbar sympathetic ganglion blocks versus epidural anesthesia. J Clin Anesth. 2000 Nov;12(7):525-30. doi: 10.1016/s0952-8180(00)00207-5. PMID 11137413
- [Background] Jo YY, Chang YJ, Kim YB, Lee S, Kwak HJ. Effect of Preoperative Forced-Air Warming on Hypothermia in Elderly Patients Undergoing Transurethral Resection of the Prostate. Urol J. 2015 Nov 14;12(5):2366-70. PMID 26571323
- [Derived] Nayebi N, Tekgul ZT, Sahinkaya HH. Effect of Prewarming on Skin Temperature Changes After Spinal Anesthesia in Transurethral Resection of the Bladder. J Perianesth Nurs. 2024 Jun;39(3):391-396. doi: 10.1016/j.jopan.2023.08.020. Epub 2024 Jan 11. PMID 38206216